CLINICAL TRIAL: NCT07378228
Title: Clinical Application and Mechanistic Study of National Traditional Chinese Medicine Master Lu Fang's "Weak Pulse at Yang and Wiry Pulse at Yin" Theory in Treating Angina Pectoris of qi Deficiency and Blood Stasis Pattern Secondary to Coronary Heart Disease
Brief Title: Weak Pulse at Yang and Wiry Pulse at Yin Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xikun Li (Other)
Responsible Party: Sponsor-Investigator, Xikun Li, Hospital Director, Harbin Traditional Chinese Medicine Hospital
Organization: Harbin Traditional Chinese Medicine Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HarbinTraditionalH
Record Dates: First submitted 2026-01-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease; Stable Angina Pectoris
MeSH Terms: conditions — Coronary Disease; Angina, Stable | interventions — Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Pharmacological Therapy (Active Comparator): Participants in this arm receive the standard pharmacological regimen for stable angina pectoris secondary to coronary heart disease. This includes oral administration of Metoprolol succinate extended-release tablets, Aspirin enteric-coated tablets, and Atorvastatin calcium tablets.
  Interventions: Drug: Metoprolol Succinate Extended-Release Tablets; Drug: Aspirin Enteric-Coated Tablets; Drug: Atorvastatin Calcium Tablets
- Conventional Therapy plus Yixin Powder (Experimental): Participants in this arm receive the same standard pharmacological regimen as the Conventional Pharmacological Therapy arm. Additionally, they receive the traditional Chinese herbal formula Yixin Powder, administered orally in divided doses.
  Interventions: Drug: Metoprolol Succinate Extended-Release Tablets; Drug: Aspirin Enteric-Coated Tablets; Drug: Atorvastatin Calcium Tablets; Drug: Yixin Powder

INTERVENTIONS:
Drug: Metoprolol Succinate Extended-Release Tablets — Metoprolol succinate extended-release tablets, 23.75 mg administered orally once daily.
Drug: Aspirin Enteric-Coated Tablets — Aspirin enteric-coated tablets, 100 mg administered orally once daily.
Drug: Atorvastatin Calcium Tablets — Atorvastatin calcium tablets, 20 mg administered orally once daily.
Drug: Yixin Powder — A traditional Chinese herbal formula composed of red ginseng (5 g), pseudo-ginseng powder (3 g), dragon's blood (1 g), leech (3 g), succinite (3 g), Chinese hawthorn fruit (10 g), and myrrh (5 g). Prepared by the hospital formulary. Administered orally at a total daily dose of 30 g, divided into two 15 g portions taken morning and evening.
  Arms: Conventional Therapy plus Yixin Powder

SUMMARY:
This is a clinical study to evaluate the effectiveness and explore the possible working mechanisms of a traditional Chinese herbal formula called Yixin Powder. The study focuses on patients with stable angina pectoris (chest pain) caused by coronary heart disease (CHD), who are diagnosed with a specific Chinese medicine pattern known as "qi deficiency and blood stasis," based on the "weak pulse at yang and wiry pulse at yin" theory.

The study hypothesizes that adding Yixin Powder to standard Western medication will be beneficial for these patients. To test this, participants diagnosed with this condition will be randomly assigned to one of two groups. One group will receive standard medication alone, while the other group will receive the same standard medication plus Yixin Powder. The effects of the treatments will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CHD-induced stable angina pectoris according to Western medicine diagnostic criteria；
* Diagnosis of qi deficiency and blood stasis pattern according to TCM pattern differentiation;
* Age between 40 and 70 years, regardless of sex;
* Stable vital signs and normal liver and renal function before enrollment;
* Angina severity graded between I and III;
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Uncontrolled severe hypertension (BP ≥180/110 mmHg);
* Severe comorbid conditions involving major organs or systems, including heart, brain, liver, or kidneys;
* Known allergy to, or intolerance of, any of the study medications; (3) Presence of psychiatric disorders;
* Requirement for long-term use of medications that could interfere with study outcomes;
* Coexisting infectious diseases.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Response Rate based on Traditional Chinese Medicine (TCM) Syndrome Score Improvement | Assessed before treatment initiation and after 4 weeks of treatment.
  The comprehensive therapeutic index (N) is calculated as: [(pre-treatment score - post-treatment score) / pre-treatment score] × 100%. Efficacy is classified as: Significant Response (N ≥ 70%), Partial Response (30% ≤ N < 70%), No Response (N < 30%), or Aggravation. The Overall Response Rate (ORR) is the proportion of participants achieving Significant or Partial Response.
Response Rate based on Electrocardiogram (ECG) Improvement | Assessed before treatment initiation and after 4 weeks of treatment.
  Efficacy is classified as: Significant Response (ECG returns to normal/near-normal), Partial Response (marked improvement in ST segments, T waves, or conduction), No Response (no significant change), or Aggravation (worsening of ECG findings). The Overall Response Rate (ORR) is the proportion of participants achieving Significant or Partial Response.

SECONDARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) Score | Assessed before treatment initiation and after 4 weeks of treatment.
  The SAQ is a disease-specific health status measure for patients with coronary artery disease. It assesses five domains: Physical Limitation, Anginal Stability, Anginal Frequency, Treatment Satisfaction, and Disease Perception. The manuscript does not specify the score range or whether a higher score indicates a better or worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xikun Li, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No